CLINICAL TRIAL: NCT01738321
Title: Changes in Intracuff Pressure of a Cuffed Endotracheal Tube During Prolonged Surgical Procedures.
Status: Completed | Type: Observational
Sponsor: Senthil G. Krishna (Other)
Responsible Party: Sponsor-Investigator, Senthil G. Krishna, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB12-00715
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiac patients: Patients undergoing cardiac surgery
  Interventions: Other: Cuff pressure
- Non-cardiac patients: Patients undergoing any surgery other than cardiac surgery
  Interventions: Other: Cuff pressure

INTERVENTIONS:
Other: Cuff pressure — Measuring endotracheal tube (ETT) cuff pressure

SUMMARY:
To date, there are no data in the literature regarding changes in the intracuff pressure during prolonged surgical procedures. It is possible that the pressure will increase over time related to gas expansion during equilibration to body temperature. If this is the case, these patients may be at risk for tracheal damage. This is a prospective study to evaluate the changes in intracuff pressure over time during prolonged surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom a cuffed endotracheal tube is to be used for surgical procedures of more than 4 hours.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery lasting longer than 4 hours.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Kako H, Alkhatib O, Krishna SG, Khan S, Naguib A, Tobias JD. Changes in intracuff pressure of a cuffed endotracheal tube during surgery for congenital heart disease using cardiopulmonary bypass. Paediatr Anaesth. 2015 Jul;25(7):705-10. doi: 10.1111/pan.12631. Epub 2015 Mar 4. PMID 25735902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Patients | Non-cardiac Patients
Started | 33 | 30
Completed | 33 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiac Patients | Non-cardiac Patients | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 30 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.8 (3.6) | 9.9 (5.1) | 8.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Intracuff Pressure
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Cardiac Patients | Non-cardiac Patients
Number analyzed (Participants) | 33 | 30
cmH2O | -11.8 (6.4) | -9.5 (29.7)

ADVERSE EVENTS:
Arm/Group | Cardiac Patients | Non-cardiac Patients
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 0/33 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes